CLINICAL TRIAL: NCT03926273
Title: Serum and Urine Ghrelin in Adult Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, rania sanad, Principal Investigator, Zagazig University
Other Study IDs: ZU-IRB#5271\ 2-6-2018
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy
Keywords: epilepsy; serum ghrelin; urine ghrelin
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Epileptic participants group consisted of 40 adults (15 females and 25 males) clinically and electrophysiological were diagnosed according to the international league against epilepsy classification 2010.
- group 2: Control group consisted of 40 adults (16 females and 24 males) non - epileptic healthy subjects.

SUMMARY:
Several neuropeptides have concerned with epilepsy pathogenesis, ghrelin showed an anticonvulsant effect. There is a potential relation between its level and antiepileptic drugs (AED) response.

DETAILED DESCRIPTION:
Several neuropeptides have concerned with epilepsy pathogenesis, ghrelin showed an anticonvulsant effect. There is a potential relation between its level and antiepileptic drugs (AED) response. Objective: to evaluate ghrelin effect in adult epileptic patients and in response to AED. Methods: This case control study included 40 adult epileptic patients and 40 healthy controls. Participants were subjected to history taking of seizure semiology, full general and neurological examination, electroencephalography and cranial CT or MRI. Fasting serum acylated ghrelin (AG) and unacylated ghrelin (UAG) and urine AG levels were estimated to all participants by enzyme - linked immunosorbent assay (ELIZA).

ELIGIBILITY:
Inclusion Criteria:

* All participants were included if their age more than or equal to 18 years. Body mass index < 30 kg/m2, total cholesterol < 200mg/dl, serum triglycerides < 200 mg/dl and random blood glucose level < 126 mg/dl.

Exclusion Criteria:

* Participants had acute or chronic metabolic disorders (liver, kidney, thyroid, endocrine or gastrointestinal disorders).
* Females with irregular menstrual cycle or on estrogen therapy (7).
* Participants with organic cerebral lesion that was detected on cranial computed tomography (CT) or cranial magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The present study was a case control type. All patients were selected from out- patient clinic of Neurology department, Zagazig university hospitals, Sharkia Governorate, Egypt in the period from July 2018 to January 2019.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Serum ghrelin in Adult Epileptic Patients | 6 months
  evaluation of the effect of Serum ghrelin in adult epileptic patients and in their response to anti- epileptic drugs
Urine ghrelin in Adult Epileptic Patients | 6 months
  evaluation of the effect of Urine ghrelin in adult epileptic patients and in their response to anti- epileptic drugs

CONTACTS AND LOCATIONS:
Overall Officials: nageeb rania, PI, Principal Investigator — zagazig U
Locations (1):
- Nageeb, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
Access Criteria: after publishing the manuscript in the Egyptian journal of neurology, psychiatry and neurosurgery
URL: http://ejnpn.springeropen.com